CLINICAL TRIAL: NCT00426972
Title: A Double Blind, Placebo Controlled Trial to Investigate the Efficacy of Zesteem (Estradiol) in Accelerating the Healing of Split Thickness Skin Graft Donor Sites.
Brief Title: Trial of Zesteem (Estradiol) in Healing of Split Thickness Skin Graft Donor Sites
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Renovo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RN1002-0066
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Burn; Trauma; Varicose Ulcer
MeSH Terms: conditions — Burns; Wounds and Injuries; Varicose Ulcer | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: estradiol (Zesteem)

SUMMARY:
This trial will assess the effects of Zesteem (estradiol) on the healing of split thickness skin graft donor sites in patients aged 18-85 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85 years who have provided written informed consent.
* Patients requiring skin grafting due to burns, trauma or chronic venous ulcers, with a donor site expected to be between 20 and 200 cm2 on a non-articulated area.
* Female patients of child bearing potential who are using method(s) of contraception acceptable to the Investigator and agree to do so from at least the screening visit until one month after administration of the final study dose.

Exclusion Criteria:

* Patients with burns involving more than 15% of their total body area.
* Patients with sepsis, haemodynamic instability requiring pressor support or positive blood microbiology cultures within 48h of surgery.
* Patients with inhalation injury requiring artificial respiratory assistance.
* Patients requiring skin grafts following removal of suspicious skin lesions.
* Patients who have received treatment with systemic steroids during the 30 days prior to surgery.
* Patients who have received immunosuppressive drugs, radiation or chemotherapy during the three months prior to surgery.
* Patients with a history of malignancy in the previous three years.
* Patients with uncontrolled diabetes or diabetic ulcers.
* Patients with diseases or conditions that could, in the opinion of the Investigator, interfere with the assessment of safety, tolerability or efficacy.
* Patients who have previously had skin grafts harvested from the area to be studied.
* Patients with a skin disorder that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial.
* Patients with a history of clinically significant hypersensitivity to any of the drugs or surgical dressings to be used in this trial.
* Patients who are taking, or have taken, any investigational drugs within 3 months prior to the screening visit.
* Patients undergoing investigations or changes in management for an existing medical condition.
* Patients who are or who become pregnant up to and including Day 0 or who are lactating.
* In the opinion of the Investigator, a patient who is not likely to complete the trial for whatever reason.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Complete wound closure of skin graft donor site.

SECONDARY OUTCOMES:
Adverse events
Skin graft take

CONTACTS AND LOCATIONS:
Overall Officials: Ken Dunn, MD, Principal Investigator — Wythenshawe Hospital
Locations (29):
- Germany (14):
  - Universitatsklinikum Aachen Klinik fur Plastiche Chirurgie, Aachen
  - Universitatsklinik fur Plastiche Chirurgie und Schwerbrandverletze, Bochum
  - Klinik fur Dermatologie und Allergologie, Bochum St Josef Hospital, Bochum
  - Klinikum Koln-Merheim Abteilung Plastiche-, Rekonstruktive-, Asthetische- Hand- Verbrennungschirurgie, Cologne
  - Carl- Thiem- klinikum Cottbus, Cottbus
  - Abteilung fur Plastiche und Handchirurgie, Erlangen
  - Zentrum der Dermatologie und Venerologie, Johann Wolfgang Institut, Frankfurt
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Klinik fur Plastiche- Hand und Wiederherstellungschirurgie, Hanover
  - Klinik fur Dermatologie, Friedrich-Schiller Universitat Jena, Jena
  - Klinikum St. Georg- Leipzig, Leipzig
  - Otto-von-Gericke Universitat Magdeburg, universitatsklinikum fur Dermatologie und Venerologie, Magdeburg
  - Klinik fur Plastiche-Asthetische- u. Handchiurgie. Kinikum Offenbach, Offenbach
  - HSK, Wilhelm Fresenius Klinik, Wiesbaden
- P Stradins Clinical University Hospital, Riga, Latvia
- Russia (8):
  - Regional Clinical Hospital, Partizana, Krasnoyarsk
  - City Clinical Hospital # 36, Moscow
  - Russian Medical Academy for Postgraduate Education, Surgery, Moscow
  - City Clinical Hospital #13, Moscow
  - The Central Clinical Hospital # 1 of LLC "Russian Railways", Moscow
  - Research Institute for Traumatology and Orthopaedy, Verhne-Volzhskaya Naberezhnaya, Novorogod
  - City Clinical Hospital # 7, Saratov
  - Clinical Hospital n.a. N.V. Solovyov, Yaroslavl
- United Kingdom (6):
  - Stoke Mandeville Hospital, Aylesbury, Buckinghamshire
  - Pinderfields Hospital, Aberford Road, Wakefield
  - McIndoe Burns Unit, Queen Victoria Hospital, East Grinstead, West Sussex
  - Selly Oak Hospital, Birmingham
  - Broomfield Hospital, Chelmsford
  - Wythenshawe Hospital, Manchester